CLINICAL TRIAL: NCT05779241
Title: A Multi Dose, Open-Label, Parallel-Group Study to Evaluate the PK and Safety/Tolerability of Long-Acting Oral Risperidone (LYN-005) in Participants With Schizophrenia or Schizoaffective Disorder
Brief Title: Study to Evaluate the Pharmacokinetics (PK) and Safety/Tolerability of Long-Acting Oral LYN-005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lyndra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYN 005-C-301
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYN-005 Containing 15-mg Risperidone (Experimental): During the run-in period (Day -7 to Day -1), participants receive Risperdal® (IR risperidone) daily. During the treatment period, participants receive 5 weekly doses of LYN-005 15 mg (Days 1, 8, 15, 22, and 29) and Risperdal 1 mg from Day 1 to Day 7.
  Interventions: Drug: LYN-005; Drug: Risperidone
- LYN-005 Containing 45-mg Risperidone (Experimental): During the run-in period (Day -7 to Day -1), participants receive Risperdal® (IR risperidone) daily. During the treatment period participants receive 5 weekly doses of LYN-005 45 mg (Days 1, 8, 15, 22, and 29) and Risperdal 3 mg from Day 1 to Day 7.
  Interventions: Drug: LYN-005; Drug: Risperidone

INTERVENTIONS:
Drug: LYN-005 — Risperidone long-acting oral capsule
Drug: Risperidone — Risperidone immediate release (IR) oral tablets
  Other Names: Risperdal

SUMMARY:
Lyndra Therapeutics, Inc. is developing LYN-005, a long-acting oral (LAO) capsule (LYNX™ dosage form) of risperidone. This pivotal study (LYN-005-C-301) will evaluate the PK as well as safety and tolerability of multiple administrations of the LYN-005 formulation at two dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 and ≤64 years.
2. Current diagnosis of schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria as confirmed by the Mini International Neuropsychiatric Interview for Psychotic Disorder Studies (MINI) version 7.0.2.
3. The following psychiatric criteria are to be used to determine participant eligibility:

   1. Duration of diagnosis of schizophrenia or schizoaffective disorder of ≥2 years.
   2. Outpatient; not hospitalized for worsening of schizophrenia within the last 6 months (partial hospitalization for social management within this time period is acceptable).
   3. Medically stable over the last month and psychiatrically stable without significant symptom exacerbation over the last 3 months.
4. Stabilized on an oral antipsychotic medication (single agent) for a minimum of 6 weeks at the time of Screening.
5. On a stable dosage of all permitted non-antipsychotic medications (except for medication to be used on an as-needed basis) for at least 1 month before the Screening visit and for the duration of the study.
6. Clinical Global Impression-Severity (CGI-S) score of ≤4 (moderately ill) at screening.
7. PANSS score of ≤80 points at screening.
8. Body mass index (BMI) ≥18 kg/m2 and ≤38 kg/m2.
9. Able to read and understand study procedures and provide written informed consent before the initiation of any protocol-specific procedures.
10. Willing to comply with all protocol-specified procedures and availability for the duration of the study.

Exclusion Criteria:

1. Participants with known clinically significant esophageal or gastrointestinal (GI) disease, including but not limited to:

   1. Known strictures such as esophageal web, pyloric stenosis, or small intestinal stricture, or participants with high risk of stricture, eg, Crohn's disease.
   2. Diagnosis of a condition known to elevate or lower gastric pH, eg, achlorhydria or hypochlorhydria.
   3. Prior varices or small or large bowel obstructions.
   4. Prior abdominal or upper gastrointestinal surgery (prior uncomplicated laparoscopic procedures including appendectomy or colectomy are permitted).
   5. History of dysphagia or aspiration in the last 5 years.
   6. History of an esophageal motility disorder or undergoing treatment for a gastric motility disorder.
   7. Significant history of diarrhea or constipation within 3 months of Screening. For constipation, 2 or more of the following in the preceding 12 months (the episodes need not be consecutive): i. Straining >1/4 of defecations; ii. Lumpy or hard stools >1/4 of defecations; iii. Sensation of incomplete evacuation >1/4 of defecations; iv. Sensation of anorectal obstruction/blockage >1/4 of defecations; v .Manual maneuvers to facilitate >1/4 of defecations (e.g., digital evacuation, support of the pelvic floor); vi.<3 defecations per week; vii. Loose stools are not present, and there are insufficient criteria for irritable bowel syndrome.
   8. Multiple episodes of abdominal pain within 3 months of Screening.
   9. Moderate or severe dysmenorrhea or menorrhagia (with use of pain medication) within 3 months of Screening.
   10. History of moderate to severe Acid Reflux Disease or a score of ≥2 on the Acid Reflux Severity Scale (ARSS) [2] , indicating moderate to severe symptoms.
2. PILL-5 questionnaire score of 5 or greater.
3. Medical history or current diagnoses indicating the presence of any of the below conditions:

   1. Presence of an uncontrolled, unstable, clinically significant medical condition that could put the participant at risk because of participation in the study, interfere with the participant's ability to participate in the study or influence the interpretation of safety or PK evaluations.
   2. History of a major cardiovascular event (myocardial infarction, cardiac surgery or revascularization, unstable angina, stroke, or transient ischemic attack) or a hospitalization for heart failure with 6 months of Screening.
   3. Any clinically significant illness, medical or surgical procedure or trauma within 4 weeks of Screening.
   4. Known immunocompromised status, including individuals who have undergone organ transplantation, on immunosuppression for an immune mediated disease, or are positive for human immunodeficiency virus (HIV).
   5. Positive test for active hepatitis B or C at Screening. Participants with successfully treated hepatitis B infection which has been resolved for greater than 1 year or successfully treated hepatitis C infection will not be excluded.
   6. Donated more than 250 mL of blood within 30 days of Screening.
   7. Have difficulties with venipuncture/cannulation, including difficulty accessing veins for blood sampling and/or history of coagulopathy or endocarditis.
   8. Current DSM-5 diagnosis of major depressive episode, panic disorder, agoraphobia, social anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder on the MINI 7.0.2 or in the judgment of the Investigator. (Note that individuals with depression secondary to schizoaffective disorder are eligible).
   9. Suicidal ideation associated with actual intent and a method or plan in the past 6 months, as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS; ie, "Yes" answers on items 4 or 5) at Screening or Day -7, or having made a suicide attempt within the last 2 years.
   10. Known or suspected (non -febrile) seizure disorder.
   11. History of neuroleptic malignant syndrome.
   12. Current or history of clinically significant tardive dyskinesia.
   13. Known or suspected diagnosis of intellectual disability or organic brain disorder or other diagnosis that is primarily responsible for current symptoms and functional impairment.
   14. Medically non-adherent in the management of their schizophrenia/schizoaffective disorder.
4. Use of the below medications/treatments in the 2 weeks before enrollment, including:

   1. Proton pump inhibitors or H2 blockers.
   2. Prokinetic agents.
   3. Medications that may interfere with the absorption, metabolism, or excretion of risperidone, e.g.: i. Drugs metabolized via cytochrome P450 3A4 (CYP3A4) pathway, such as macrolide antibiotics and azole antifungals); ii. Moderate or strong CYP3A4 p-glycoprotein enzyme inducers and inhibitors (carbamazepine, phenytoin, rifampicin, phenobarbital, itraconazole, verapamil); iii. Moderate or strong cytochrome P450 2D6 (CYP2D6) inhibitors (e.g., fluoxetine, fluoxetine combinations, paroxetine, or quinidine).
   4. Concomitant medications, natural remedies, supplements, or vitamins which are associated with changes to gastric motility or pH. Use of antacids is permissible, except within 2 hours of dosing with LYN-005.
   5. Use of more than one antidepressant; or if on just one, a change in dose within 6 weeks of Screening.
   6. Depot antipsychotic use within 9 months of Screening.
   7. Electroconvulsive therapy within 3 months of Screening.
5. Participants with clinically significant abnormal safety (e.g. physical examination, vital sign) or safety laboratory assessments, specifically:

   1. Presence of a clinically significant abnormal laboratory result on blood or urine safety tests at Screening.
   2. Anemia (hemoglobin below lower limit of normal reference range) at Screening.
   3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≥3.0 × upper limit of normal (ULN), or total bilirubin ≥1.5 × ULN.
   4. Moderate or severe renal insufficiency at Screening (glomerular filtration rate <60 mL/min, as determined using the Cockcroft-Gault formula).
   5. Heart rate <50 beats per minute (bpm).
   6. Systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg at Screening.
   7. Orthostatic hypotension (or history of orthostatic hypotension), defined as a decrease of ≥20 millimeters of mercury (mmHg) in systolic pressure or a decrease of ≥10 mm Hg in diastolic pressure after 2 minutes of standing, or if standing causes signs and symptoms, at Screening or Day -7
   8. Glycated hemoglobin (HbA1c) ≥7.0%.
   9. Positive fecal occult blood test.
   10. Clinically significant prolactin elevation (≥200 ng/mL for females; ≥100 ng/mL for males).
6. Participants with the below specified patterns of substance use :

   1. Fulfillment of the DSM-5 criteria for moderate or severe substance use disorder (excluding nicotine and caffeine) within 6 months of Screening.
   2. History of alcohol consumption exceeding moderate use; in males exceeding 21 units per week and in females exceeding 14 units per week (1 unit = 360 ml beer, 25 mL of 40% spirit or 125 mL wine) over the past month. Participants are not permitted to consume alcohol during the inpatient stay nor 12 hours before any clinic visit while outpatient.
   3. Positive ethanol breathalyzer at Screening or Day -7.
   4. Positive urine drug screen for substances of abuse other than cannabis at Screening or Day -7.
   5. Heavy nicotine use (consumption of >40 cigarettes or >36 mg of nicotine from other sources [eg, vaping products] daily) or daily use of smokeless tobacco.
7. Participants of reproductive potential who are (hetero) sexually active but unwilling to use acceptable means of contraception through the Safety Follow-up (SFU). For clarity, participants who are at least 1 year post-menopausal are not of reproductive potential. Acceptable means of contraception include:

   1. Participants who have been surgically sterilized (males who have undergone a vasectomy at least 3 months before LYN-005 and have a documented negative sperm count test; females who have undergone tubal ligation or hysterectomy).
   2. Females of reproductive potential: diaphragm, injectable, oral/patch contraceptives for a minimum of 6 weeks, contraceptive sponge, implant, or intrauterine device in use before enrollment.
   3. Males: condom in combination with any of the above means of contraception.
   4. All participants: abstinence may be an acceptable means of contraception as long as the individual consents to initiate immediate use of double barrier protection for the duration of the study should (hetero) sexual intercourse occur.
8. Participants who are nursing or who have positive or indeterminate pregnancy tests at either Screening (serum test) or Day -7 (urine test).
9. Use of any experimental agent within 1 month or 5 half-lives of Screening, whichever is longer.
10. Participants who are employees or immediate family members of employees of the site, Sponsor or study-related vendors.
11. History of a serious allergic or hypersensitivity reaction to risperidone or LYN-005 excipients (refer to Investigator's Brochure).
12. Participants with history of X-ray, computed tomography scan or angiogram of the abdomen within one year of Screening.
13. Participants with CYP2D6 poor or underdetermined metabolizer status based on genetic testing.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Minimum Observed Concentration (Cmin) at Week 1 | up to Day 36
Minimum Observed Concentration (Cmin) at Week 5 | up to Day 36
Maximal Observed Concentration (Cmax) at Week 5 | up to Day 36
Average Concentration Over the Dosing Interval (Cavg) at Week 5 | up to Day 36

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) From Week 1 to Week 5 | Week 1 to Week 5
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) to Week 5 | Baseline, up to Week 5
  The total score range for the PANSS is 30-210. Higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Scranton, MD, MPH, Principal Investigator — Lyndra Therapeutics INC
Locations (5):
- United States (5):
  - CenExel CNS, Garden Grove, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Hassman Research Institute, Marlton, New Jersey
  - Community Clinical Research, Inc., Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Citrome L, Nagaraj N, Traverso G, Dumas T, Scranton R. Long-acting oral weekly risperidone (LYN-005) for schizophrenia in the USA (STARLYNG-1): a multicentre, open-label, non-randomised phase 3 trial. Lancet Psychiatry. 2025 Jul;12(7):504-512. doi: 10.1016/S2215-0366(25)00135-X. PMID 40506209